CLINICAL TRIAL: NCT06810739
Title: A Hybrid Type III Effectiveness - Implementation, Pragmatic Intervention Trial for Cervical Cancer Screen and Treat in Mozambique
Brief Title: The Women's Screening and Self-Testing Program (PROMETA) Study
Acronym: PROMETA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-1641; U01CA294674 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Human Papilloma Virus Related Cervical Carcinoma
Keywords: Human Immunodeficiency Virus; Self swab; Mozambique; Cervical cancer; Implementation science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV DNA testing from self-collected vaginal swab (Experimental): After providing informed consent, the study clinician will open a Case Report Form (CRF) for each patient which starts with a brief questionnaire which will include the participant's demographic information and medical history, including HIV viral load and CD4 counts, previous cervical cancer screening results if previously screened, and result of rapid pregnancy test performed that day with a urine sample. Each participant will then be accompanied to a private location where the study nurse will provide counseling and instruction on how to appropriately perform the self-collection vaginal swab technique. Data on HPV testing, VAT results, and referrals along each step of the process will be documented in the CRF.
  Interventions: Diagnostic Test: HPV DNA testing be self-collected vaginal swab

INTERVENTIONS:
Diagnostic Test: HPV DNA testing be self-collected vaginal swab — Directly following collection of the vaginal self-swab sample, the participant will be taken back to the waiting area and her sample will be taken to the laboratory for HPV testing using the Xpert HPV Test on the GeneXpert platform (Cepheid, Sunnyvale, CA, USA). This point-of-care test takes approximately 45 minutes to get results.

SUMMARY:
This proposal directly addresses the ability to safely scale-up a Screen-Triage-Treat approach to cervical cancer screening. The investigators propose to capitalize on a pool of screen-eligible women accessing routine care within targeted human immunodeficiency virus (HIV) care and treatment services. The primary outcome of interest is the number of women screened and the proportion of screen-positive women undergoing treatment. Secondary outcomes will focus on other implementation outcomes, and if successful, will be utilized to inform future research to take this approach to scale across Mozambique.

DETAILED DESCRIPTION:
This study will use a hybrid type III effectiveness-implementation design. In a hybrid type III design, the primary focus is on testing of an implementation strategy, while simultaneously continuing to observe and gather information on the effectiveness of a clinical intervention, under real world conditions, for which effectiveness data has already largely been determined. Best practices for deploying the Screen-Triage-Treat approach to cervical cancer screening utilizing self-collected human papilloma virus (HPV) deoxyribonucleic acid (DNA) testing within Mozambique´s HIV care and treatment services will be evaluated. The study will employ a mixed-methods approach, collecting both quantitative and qualitative data. The primary outcome of interest is the number of women screened and the proportion of HPV screen-positive women undergoing treatment, while secondary outcomes will focus on other implementation outcomes, and if successful, will be utilized to inform future research to take this approach to scale across Mozambique.

ELIGIBILITY:
Inclusion Criteria:

* Women 25-49 years
* Accessing HIV care and treatment services
* Not being pregnant
* Patients with a cervix

Exclusion Criteria:

* Physical or mental impairment that inhibits participation in the study
* Pregnant women or <6 weeks post-partum
* Women who have undergone a total hysterectomy with removal of the cervix

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 8445 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The number of women screened and the proportion of screen-positive women successfully undergoing treatment or evaluation/referral. | 2.5 Years
  Baseline data will be retrospectively collected for the prior 12 months at each of the selected study sites, including the number of women accessing care for HIV care and treatment services each month; the number of women screened for cervical cancer through standard of care protocols; the proportion of screen-positive women who then received treatment or referral for treatment, and the length of time between screening positive and receiving treatment if appropriate.

SECONDARY OUTCOMES:
Test Result Notification Rate | 2.5 Years
  The proportion of women who were notified of their HPV DNA test result on the same day as sample collection.
Treatment Rate | 2.5 Years
  The proportion of screen-positive women who were treated with thermal ablation, if appropriate, or referred for higher level of care or return appointment.

CONTACTS AND LOCATIONS:
Overall Officials: D. Troy Moon, MD, MPH, Principal Investigator — Tulane University
Locations (1):
- University Eduardo Mondlane (UEM), Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon TD, Salcedo MP, Mavume-Mangunyane E, Sidat M, Lorenzoni C, Baker E, Amorim G, Paz-Soldan VA, Kampa KT, Condon K, Myers H, Sacarlal J. A hybrid type III effectiveness-implementation study designed to test implementation best practices of deploying a Screen-Triage-Treat approach to cervical cancer screening and management utilizing self-collected HPV DNA testing in Chokwe District, Mozambique. BMC Public Health. 2025 Nov 25;26(1):6. doi: 10.1186/s12889-025-25730-5. PMID 41291606